CLINICAL TRIAL: NCT04121741
Title: Evaluating the Impact of Singing Interventions on Markers of Cardiovascular Health in Older Patients With Cardiovascular Disease
Brief Title: Singing and Cardiovascular Health in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jacquelyn Kulinski, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 35864; R33AT010680 (NIH)
Record Dates: First submitted 2019-10-07; First posted 2019-10-10 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor; Cardiovascular Health
Keywords: Singing
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Singing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Singing intervention 1 (Active Comparator): Instructional sing-a-long video. A video series will be created and recorded for the purposes of the study. Flow Mediated dilation (FMD) and EndoPAT will be measured before and after singing.
  Interventions: Other: Singing with Guided Video
- Singing intervention 2 (Active Comparator): In-person music therapy session. The music therapist will continue to coach throughout the 30-minute session. Flow Mediated dilation (FMD) and EndoPAT will be measured before and after singing.
  Interventions: Other: Singing with Music Therapist
- Control/sham intervention (Sham Comparator): Subjects will have a 30-minute period of rest sitting upright (as they would be positioned for the singing interventions). This arm is meant to isolate the specific effects of the treatment rather than the potential "incidental" effects related to the research setting and measurements. During this time, subjects will undergo hearing testing. Flow Mediated dilation (FMD) and EndoPAT will be measured before and after the 30 minute rest.
  Interventions: Other: Control Arm

INTERVENTIONS:
Other: Singing with Music Therapist — Music therapy sessions will begin with vocal and breathing warm-up exercises for about 10 minutes. The Music Therapist will play the songs (chosen from a list by the subject) to sing along to and will alter the characteristics of the music (volume, tempo, level of support) to ensure a successful experience for subjects and motivate them to put forth more effort into singing the song. The music therapist will continue to coach throughout the 30-minute session, reminding subjects of strategies practiced and how to implement those strategies while singing. Music therapy sessions will be led by Erica Flores, MT-BC, WMTR, Owner of Healing Harmonies Music Therapy, or a member of her team. Erica and her team of MTs were trained in Neurological Music Therapy.
  Arms: Singing intervention 2
Other: Singing with Guided Video — The videos will include a vocal warm-up (10 minutes long). The subject will then have the option to select and sing two songs (10 minutes each), with offerings in four music genres including Folk, Pop, Country, and a Hymn. Each piece will vary in tempo, melodic contour, and rhythm. The total duration of singing via this format will be 30 minutes.
  Arms: Singing intervention 1
Other: Control Arm — 30 minute rest period, no singing will take place during this arm. During this rest period a member of the study team will assist the subject in a hearing test using headphones, a tablet, and a trumpet app. This is done to asses the current hearing level of the subject.
  Arms: Control/sham intervention

SUMMARY:
Cardiovascular disease (CVD) claims more lives each year than cancer and chronic respiratory disease combined. Participation in cardiac rehabilitation (CR) reduces mortality and risk of a major cardiovascular event in secondary prevention populations, including older adults. Older adults are less likely to participate in CR, as comorbidities in this population, including arthritis and chronic obstructive pulmonary disease, make participation difficult. Singing is a physical activity that involves components of the vagal nerves manifested as changes in cardiac autonomic regulation. Unlike physical exercise, the effects of singing on cardiovascular health has not been well-studied. The hypothesis for this project is that older patients with CVD will have favorable improvement in cardiovascular biomarkers, including, endothelial function and heart rate variability (HRV), after 30 minutes of singing.

DETAILED DESCRIPTION:
This proposal seeks to create, optimize and test two different singing interventions in older patients with CVD. The study will consist of three arms, according to a randomized, single-blind, crossover, sham procedure-controlled design. Sixty-five total participants will each have three visits on three different occasions for the following interventions:

1. a 30-minute period of guided singing from an in-person music therapist
2. a 30-minute period of singing along to an instructional video including a professor of voice and "inexperienced, older singing student"
3. a 30-minute sham intervention (subjects will undergo a hearing test)

The goal will be to determine which singing intervention, if any, is superior to the other - as this would be important to guide longer and larger clinical trials in the field. Knowledge gained from this proposal will improve understanding of biologic mechanisms of singing behaviors, as it relates to CVD.

ELIGIBILITY:
Inclusion Criteria:

* English Speaking
* Have a history of coronary artery disease (defined as history of myocardial infarction, coronary stenosis >50%, percutaneous coronary intervention with stent placement, balloon angioplasty, or coronary arterial bypass grafting)

Exclusion Criteria:

* Subjects with a permanent pacemaker or implantable cardioverter defibrillator (ICD) implanted
* Patients with a history of atrial fibrillation, flutter or atrial tachycardia
* Parkinson's disease or a tremor
* Amputated upper extremity or presence of upper-arm (dialysis) fistula
* Fingernail onychomycosis (fungal infections resulting in thickening of the nails)
* Pregnancy
* Current illicit drug use (marijuana, tobacco, cocaine, amphetamines, etc.)
* Current excessive alcohol use (defined as more than 14 drinks/week for women, more than 28 drinks/week for men)
* Unstable coronary heart disease (active symptoms of chest discomfort)
* History of a Stroke or TIA or peripheral arterial disease
* Known history of cognitive impairment or inability to follow study procedures
* Cancer requiring systemic treatment within five years of enrollment.
* Subjects requiring supplemental oxygen use
* Non-English speaking subjects (video with lyrics are taped in English)

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Derived] Bagherimohamadipour M, Hammad M, Visotcky A, Sparapani R, Kulinski J. Effects of singing on vascular health in older adults with coronary artery disease: a randomized, crossover trial. Front Cardiovasc Med. 2025 Apr 28;12:1546462. doi: 10.3389/fcvm.2025.1546462. eCollection 2025. PMID 40357442
- [Derived] Bagherimohamadipour M, Hammad M, Visotcky A, Sparapani R, Kulinski J. Effects of Singing on Vascular Health in Older Adults with Coronary Artery Disease: A Randomized Trial. medRxiv [Preprint]. 2024 Jul 27:2024.07.25.24311033. doi: 10.1101/2024.07.25.24311033. PMID 39108506

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in January of 2020 and concluded in August 2023 as enrollment goals were met successfully. Subjects were identified by reviewing the electronic medical records of patients visiting the outpatient clinic. Subjects were also identified using a cohort discovery tool from the institution's Clinical Research Data Warehouse.
Pre-assignment Details: Randomized, single-blind, crossover, sham procedure-controlled design. Each subject will have 3 visits: (1) a 30-minute period of guided singing from a music therapist, (2) a 30-minute period of singing along to an instructional video (3) a 30-minute rest period without any intervention. There will be a washout period between visits of a minimum of 2 days and a maximum of 7 days (to allow for wash-out effects of the prior intervention). Visits are coded ABC. A-Control, B-Coach, C-video
Groups:
- Randomization ABC; Randomization ACB; Randomization BAC; Randomization BCA; Randomization CAB; Randomization CBA: A- Control B- Singing Intervention with Coach C- Singing Intervention with Sing-a-long Video
  Control Visit: 30 minute rest period, no singing will take place during this arm. This arm is meant to isolate the specific effects of the treatment rather than the potential "incidental" effects related to the research setting and measurements. During this time, subjects will undergo hearing testing.
  Singing with Music Therapist: Music therapy sessions will begin with vocal and breathing warm-up exercises for about 10 minutes. The Music Therapist will play the songs (chosen from a list by the subject) to sing along to and will alter the characteristics of the music (volume, tempo, level of support) to ensure a successful experience for subjects and motivate them to put forth more effort into singing the song. The music therapist will continue to coach throughout the 30-minute session, reminding subjects of strategies practiced and how to implement those strategies while singing.
  Instructional sing-a-long video. A video series will be created and recorded for the purposes of the study. The videos will include a vocal warm-up (10 minutes long). The subject will then have the option to select and sing two songs (10 minutes each), with offerings in four music genres including Folk, Pop, Country, and a Hymn. Each piece will vary in tempo, melodic contour, and rhythm. The total duration of singing via this format will be 30 minutes.
Period: Overall Study
Arm/Group | Randomization ABC | Randomization ACB | Randomization BAC | Randomization BCA | Randomization CAB | Randomization CBA
Started | 11 | 11 | 10 | 11 | 11 | 11
Completed | 10 | 11 | 10 | 11 | 11 | 11
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible subjects must be English speaking, between the ages of 55-79 years, have a history of coronary artery disease (defined as history of myocardial infarction, coronary stenosis >50%, percutaneous coronary intervention with stent placement, balloon angioplasty, or coronary arterial bypass grafting).
Groups:
- Entire Study Population: All 65 participants who signed informed consent and participated in this study.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 65
Age, Customized [Median (Full Range); unit: years]
  Age at Screening | 68.2 [55.1 to 78.7]
Age, Customized [Mean (Full Range); unit: years]
  Age at Screening | 67.7 [55.1 to 78.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 64
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 56
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 65
History of Heart Attack (Myocardial Infarction) [Number; unit: participants] | 41
History of Stent Placement [Number; unit: participants] | 47
History of Coronary Artery Bypass (CABG) [Number; unit: participants] | 18
History of Diabetes Mellitus [Number; unit: participants] | 19
History of Hypertension [Number; unit: participants] | 49
History of High Cholesterol [Number; unit: participants] | 55
History of Chronic Kidney Disease [Number; unit: participants] | 10
History of Respiratory Illness [Number; unit: participants] | 18
History of Past Smoking [Number; unit: participants] | 26
History of Heart Failure [Number; unit: participants] | 12
Body Mass Index (BMI) Category [Number; unit: participants]
  Underweight <18.5 | 4
  Healthy weight 18.5 - 24.9 | 12
  Overweight 25 to 29.9 | 17
  Obese 30 or greater | 32
Godin Category [Number; unit: participants]
  Less than 14 Insufficiently Active | 10
  14-23 Moderately Active | 10
  24 or more Active | 45
Hearing Test Results - Left Ear [Number; unit: participants] — Population: One subject was unable to get a hearing test performed during the study procedures as the app that was used to perform the test malfunctioned and would not open due to needing an update.
  participants
    Normal: number analyzed (Participants) | 64
    Normal | 20
    Mild Loss: number analyzed (Participants) | 64
    Mild Loss | 14
    Moderate Loss: number analyzed (Participants) | 64
    Moderate Loss | 22
    Severe Loss: number analyzed (Participants) | 64
    Severe Loss | 8
Hearing Test Results - Right Ear [Number; unit: participants] — Population: One subject was unable to get a hearing test performed during the study procedures as the app that was used to perform the test malfunctioned and would not open due to needing an update.
  participants
    Normal: number analyzed (Participants) | 64
    Normal | 22
    Mild Loss: number analyzed (Participants) | 64
    Mild Loss | 8
    Moderate Loss: number analyzed (Participants) | 64
    Moderate Loss | 25
    Severe Loss: number analyzed (Participants) | 64
    Severe Loss | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in FMD%
Description: Assess macrovascular endothelial function by assessing changes in post-intervention to pre-intervention changes in brachial artery FMD%.
Time Frame: At baseline and after 30-minute singing and control intervention(s)
Population: Poor quality FMD measurements were excluded from the analysis
Measure: Mean (Standard Error); unit: FMD percent
Arm/Group | Singing Intervention 1 | Singing Intervention 2 | Control/Sham Intervention
Number analyzed (Participants) | 63 | 62 | 61
FMD percent | -0.06 (0.30) | -0.11 (0.31) | -0.06 (0.31)
Statistical Analysis 1: Comparison: Singing Intervention 1 vs Control/Sham Intervention; Test type: Superiority; p = 0.864, Regression, Linear — Using Bonferroni correction for 3 primary outcomes (FMD, RHI, fRHI), a priori threshold for statistical significance was p<0.0167; Included outlier detection and removal with estimation of standard models for a three-treatment, cross-over design; Mean Difference (Final Values) = -0.07, Standard Error of Mean 0.42 — Estimated mean difference for FMD% (singing video intervention compared to control) is shown. Estimates of FMD% for singing coach intervention compared to control also performed; Please reference the following pre-print manuscript for additional statistical analyses. Bagherimohamadipour M, Hammad M, Visotcky A, Sparapani R, Kulinski J. Effects of Singing on Vascular Health in Older Adults with Coronary Artery Disease: A Randomized Trial. medRxiv [Preprint]. 2024 Jul 27:2024.07.25.24311033. doi: 10.1101/2024.07.25.24311033. PMID: 39108506; PMCID: PMC11302710
Statistical Analysis 2: Comparison: Singing Intervention 2 vs Control/Sham Intervention; Test type: Superiority; p = 0.913, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Included outlier detection and removal with estimation of standard models for a three-treatment, cross-over design; Mean Difference (Final Values) = -0.05, Standard Error of Mean 0.42 — Estimated mean difference for FMD% (singing coach intervention compared to control) is shown. Estimates of FMD% for singing video intervention compared to control also performed; [other analysis details as in outcome 1, analysis 1]

2. Primary Outcome: Change in Reactive Hyperemia Index (RHI)
Description: Assess microvascular endothelial function by measuring changes in reactive hyperemia index through finger plethysmography using EndoPAT. A larger post-intervention to pre-intervention change in RHI is considered a better outcome.
Time Frame: At baseline and after 30-minute singing and control intervention(s)
Population: Poor quality EndoPAT measurements were excluded from the analysis
Measure: Mean (Standard Error); unit: Index
Arm/Group | Singing Intervention 1 | Singing Intervention 2 | Control/Sham Intervention
Number analyzed (Participants) | 50 | 57 | 54
Index | 0.22 (0.10) | 0.19 (0.11) | 0.12 (0.09)
Statistical Analysis 1: Comparison: Singing Intervention 1 vs Control/Sham Intervention; Test type: Superiority; p = 0.290, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Included outlier detection and removal with estimation of standard models for a three-treatment, cross-over design; Mean Difference (Final Values) = 0.13, Standard Error of Mean 0.13 — Estimated mean difference for RHI (singing video intervention compared to control) is shown. Estimates of RHI for singing coach intervention compared to control also performed; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Singing Intervention 2 vs Control/Sham Intervention; Test type: Superiority; p = 0.462, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Included outlier detection and removal with estimation of standard models for a three-treatment, cross-over design; Mean Difference (Final Values) = 0.09, Standard Error of Mean 0.12 — Estimated mean difference for RHI (singing coach intervention compared to control) is shown. Estimates of RHI for singing video intervention compared to control also performed; [other analysis details as in outcome 1, analysis 1]

3. Primary Outcome: Change in Framingham Reactive Hyperemia Index (fRHI)
Description: Assess microvascular endothelial function by measuring changes in Framingham reactive hyperemia index through finger plethysmography using EndoPAT. A larger post-intervention to pre-intervention change in fRHI is considered a better outcome.
Time Frame: At baseline and after 30-minute singing and control intervention(s)
Population: Poor quality EndoPAT measurements were excluded from the analysis
Measure: Mean (Standard Error); unit: Index
Arm/Group | Singing Intervention 1 | Singing Intervention 2 | Control/Sham Intervention
Number analyzed (Participants) | 50 | 55 | 55
Index | 0.8 (0.1) | 0.6 (0.1) | 0.6 (0.1)
Statistical Analysis 1: Comparison: Singing Intervention 1 vs Control/Sham Intervention; Test type: Superiority; p = 0.005, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Included outlier detection and removal with estimation of standard models for a three-treatment, cross-over design; Mean Difference (Final Values) = 0.54, Standard Error of Mean 0.19 — Estimated mean difference for fRHI (singing video intervention compared to control) is shown. Estimates of fRHI for singing coach intervention compared to control also performed; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Singing Intervention 1 vs Control/Sham Intervention; Test type: Superiority; p = 0.570, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Included outlier detection and removal with estimation of standard models for a three-treatment, cross-over design; Mean Difference (Final Values) = 0.11, Standard Error of Mean 0.18 — Estimated mean difference for fRHI (singing coach intervention compared to control) is shown. Estimates of fRHI for singing video intervention compared to control also performed; [other analysis details as in outcome 1, analysis 1]

4. Secondary Outcome: BORG Rating of Perceived Exertion
Description: The BORG RPE scale assesses an individual's perceived level of exertion. It ranges from 6 to 20, whereas 6 reflects no exertion at all and 20 reflects maximal exertion.
Time Frame: after 30-minute singing (and sham) interventions
Population: One participant who did not complete all three interventions was not included in final analysis
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Singing Intervention 1 | Singing Intervention 2 | Control/Sham Intervention
Number analyzed (Participants) | 64 | 64 | 64
Units on a scale | 9.98 (0.28) | 10.66 (0.29) | 6.33 (0.10)

5. Secondary Outcome: Change in SDNN (Standard Deviation of Normal-to-Normal Intervals)
Description: Heart rate variability is assessed using SDNN (Standard Deviation of Normal-to-Normal intervals) before, during, and post-intervention. Reported as percent change compared to the baseline (pre) value. Percent change calculated as 100*[(post-pre)/pre] or 100*[(during-pre)/pre].
  An appropriately sized (Bluetooth-capable) chest strap (Polar, Kempele, Finland) with a heart rate sensor was applied to the subject's bare chest. Three-minute-long HRV recordings were obtained before, during, and after singing (or rest control).
Time Frame: at baseline (pre), during, and after (post) 30-minute singing and sham intervention(s)
Population: One participant who did not complete all three interventions was not included in final analysis
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Singing Intervention 1 | Singing Intervention 2 | Control/Sham Intervention
Number analyzed (Participants) | 64 | 64 | 64
percent change
  (Post-Pre) SDNN Relative Difference % | 20.7 (9.7) | 22.4 (12.8) | 29.5 (22.5)
  (During-Pre) SDNN Relative Difference % | 14.5 (9.7) | 23.0 (21.1) | 9.2 (7.1)

6. Secondary Outcome: Change in RMSSD (Root Mean Square of Successive Differences)
Description: Heart rate variability is assessed using (RMSSD) root mean square of successive differences before, during, and post-intervention. Reported as percent change compared to the baseline (pre) value. Percent change calculated as 100*[(post-pre)/pre] or 100*[(during-pre)/pre].
  An appropriately sized (Bluetooth-capable) chest strap (Polar, Kempele, Finland) with a heart rate sensor was applied to the subject's bare chest. Three-minute-long HRV recordings were obtained before, during, and after singing (or rest control).
Time Frame: at baseline (pre), during, and after (post) 30-minute singing and sham intervention(s)
Population: One participant who did not complete all three interventions was not included in final analysis
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Singing Intervention 1 | Singing Intervention 2 | Control/Sham Intervention
Number analyzed (Participants) | 64 | 64 | 64
percent change
  (Post-Pre) RMSSD Relative Difference % | 56.9 (41.5) | 49.5 (38.9) | 62.6 (28.0)
  (During-Pre) RMSSD Relative Difference % | 52.5 (27.3) | 80.2 (57.3) | 40.6 (13.1)

7. Secondary Outcome: Change in HF Power (High-frequency Power)
Description: Heart rate variability is assessed using high-frequency power (HF Power) before, during and post-intervention. Reported as an absolute change or difference compared to baseline (pre). Unit of measurement is milliseconds-squared. Power in the High Frequency band of the HRV spectrum falls between 0.15-0.40 Hz. The actual activity in that band is typically expressed in terms of "power", which uses the units of milliseconds-squared for a particular Hertz (Hz) band. Think of it as an "area under the curve".
  An appropriately sized (Bluetooth-capable) chest strap (Polar, Kempele, Finland) with a heart rate sensor was applied to the subject's bare chest. Three-minute-long HRV recordings were obtained before, during, and after singing (or rest control).
Time Frame: at baseline (pre), during, and after (post) 30-minute singing and sham intervention(s)
Population: One participant who did not complete all three interventions was not included in final analysis
Measure: Mean (Standard Error); unit: milliseconds-squared
Arm/Group | Singing Intervention 1 | Singing Intervention 2 | Control/Sham Intervention
Number analyzed (Participants) | 64 | 64 | 64
milliseconds-squared
  (Post-Pre) HF Power Absolute Difference | 477.5 (346.3) | -334.7 (350.4) | 401.0 (203.5)
  (During-Pre) HF Power Absolute Difference | 242.7 (261.9) | -141.3 (447.1) | 423.7 (200.1)

8. Secondary Outcome: Change in LF Power (Low-frequency Power)
Description: Heart rate variability is assessed using low-frequency power (LF Power) before, during and post-intervention. Reported as an absolute change or difference compared to baseline (pre). Unit of measurement is milliseconds-squared. Power in the Low Frequency band of the HRV spectrum is defined as greater than 0.00 Hz and less than 0.04 Hz. The actual activity in that band is typically expressed in terms of "power", which uses the units of milliseconds-squared for a particular Hertz (Hz) band. Think of it as an "area under the curve".
  An appropriately sized (Bluetooth-capable) chest strap (Polar, Kempele, Finland) with a heart rate sensor was applied to the subject's bare chest. Three-minute-long HRV recordings were obtained before, during, and after singing (or rest control).
Time Frame: at baseline (pre), during, and after (post) 30-minute singing and sham intervention(s)
Population: One participant who did not complete all three interventions was not included in final analysis
Measure: Mean (Standard Error); unit: milliseconds-squared
Arm/Group | Singing Intervention 1 | Singing Intervention 2 | Control/Sham Intervention
Number analyzed (Participants) | 64 | 64 | 64
milliseconds-squared
  (Post-Pre) LF Power Absolute Difference | 1318.8 (693.9) | 636.2 (399.9) | 244.8 (350.8)
  (During-Pre) LF Power Absolute Difference | 525.3 (547.9) | 254.1 (452.0) | -19.7 (191.5)

9. Secondary Outcome: Change in LF/HF Ratio (Low-frequency to High-frequency Ratio)
Description: Heart rate variability is assessed using LF/HF ratio before, during and post-intervention. This is an (absolute) difference between ratios, so there are no units of measure.
  The LF/HF ratio is as an index of sympatho-vagal balance between the sympathetic and parasympathetic nervous systems.
  An appropriately sized (Bluetooth-capable) chest strap (Polar, Kempele, Finland) with a heart rate sensor was applied to the subject's bare chest. Three-minute-long HRV recordings were obtained before, during, and after singing (or rest control).
Time Frame: at baseline (pre), during, and after (post) 30-minute singing and sham intervention(s)
Population: One participant who did not complete all three interventions was not included in final analysis
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | Singing Intervention 1 | Singing Intervention 2 | Control/Sham Intervention
Number analyzed (Participants) | 64 | 64 | 64
Ratio
  (Post-Pre) LF/HF Ratio Absolute Difference | 0.6 (0.4) | 0.3 (0.5) | -1.0 (0.6)
  (During-Pre) LF/HF Ratio Absolute Difference | 2.2 (1.2) | -0.2 (0.7) | -0.6 (0.4)

10. Secondary Outcome: Change in LnHF Power (Natural Log (Milliseconds Squared))
Description: Heart rate variability is assessed using LnHF Power before, during and post-intervention. The physiological range for the LnHF Power in heart rate variability is typically considered to be between 4 and 7. Reported here as an absolute change or difference in LnHF Power (natural log (milliseconds squared)). Under controlled conditions while breathing at normal rates, we can use LnHF Power to estimate vagal tone.
  Interpreting results:
  Higher natural log HF power: Indicates greater parasympathetic activity, often associated with relaxation and a healthy stress response.
  Lower natural log HF power: May suggest decreased parasympathetic activity, potentially related to stress or other physiological factors.
  An appropriately sized (Bluetooth-capable) chest strap (Polar, Kempele, Finland) with a heart rate sensor was applied to the subject's bare chest. Three-minute-long HRV recordings were obtained before, during, and after singing (or rest control).
Time Frame: at baseline (pre), during, and after (post) 30-minute singing and sham intervention(s)
Population: One participant who did not complete all three interventions was not included in final analysis
Measure: Mean (Standard Error); unit: natural log (milliseconds-squared)
Arm/Group | Singing Intervention 1 | Singing Intervention 2 | Control/Sham Intervention
Number analyzed (Participants) | 64 | 64 | 64
natural log (milliseconds-squared)
  (Post-Pre) LnHF Power Absolute Change | 0.1 (0.2) | -0.2 (0.2) | 0.3 (0.2)
  (During-Pre) LnHF Power Absolute Change | -0.1 (0.2) | -0.0 (0.2) | 0.3 (0.2)

11. Other Pre Specified Outcome: Change in TNF-alpha, IL-1 Beta, IL-6, and IL-8
Description: measure the change in TNF-alpha, IL-1 Beta, IL-6, and IL-8
Time Frame: at baseline and 30 minutes later (after interventions or sham)
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Visual Mood Score
Description: Arts Observation Scale to evaluate the effect of performing arts activities in healthcare settings. Two reactions (relaxation and distraction) will be scored by the research coordinator nurse based on direct observation of the subjects during the singing intervention. The qualitative portion of this instrument enables the collection of personal feedback and quotations from subjects. Observers (research team) can also gather more detailed accounts of subjects' responses to activities, including experience and perceptions
Time Frame: at baseline and 30 minutes later (after interventions or sham)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) will be recorded with start dates occurring any time after informed consent is obtained until 7 (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation. Events will be followed for outcome information until resolution or stabilization. All serious adverse events will be promptly reported to the IRB upon awareness of the events (no longer than 24hrs after event). AEs are reported to the IRB at the annual report.
Description: For all adverse events, we will determine severity (mild, moderate, severe) and relationship, if any, to the protocol (unrelated, possibly related, or definitely related). The PI will be informed of all serious adverse events as soon as they occur.
Groups:
- Singing Intervention 1: Singing Video Intervention 30 minutes
- Singing Intervention 2: Singing Coach Intervention 30 minutes
- Control: Rest Period 30 minutes
Arm/Group | Singing Intervention 1 | Singing Intervention 2 | Control
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/65 | 0/65
Other Adverse Events (participants affected / at risk) | 0/65 | 0/65 | 2/65
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Singing Intervention 1 (N=65) | Singing Intervention 2 (N=65) | Control (N=65)
Adverse Event - Internal, Mild, Expected, Definitely Related to the Protocol (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Following FMD, subject's arm was red, painless. PI advised to not perform second FMD. Resolved spontaneously.
Adverse Event - Internal, Moderate, Unexpected, Unrelated to the Protocol (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Subject came into study visit and blood pressure was elevated by the end of the study visit. PI was notified and subject left to seek medical care. Subject's blood pressure normalized and testing was normal, no interventions were needed.

LIMITATIONS AND CAVEATS:
1. Due to technical issues related to image quality, machine/equipment malfunctions, and/or too much patient movement/patient related signal interference during testing, not all of the FMD, EndoPAT, and heart rate variability tests were included or analyzed in the final data set.
2. Due to the COVID-19 pandemic, 20 out of 64 coaching intervention visits were conducted by the singing coach remotely (via Microsoft teams) to limit any exposure for study staff and research subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT04121741/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT04121741/SAP_001.pdf
  • Informed Consent Form (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT04121741/ICF_002.pdf